CLINICAL TRIAL: NCT04358107
Title: Retrospective Study of Optimal Methods of Disease Progression and Survival Analysis in Children and Adults Patients With Adrenocortical Cancer (ACC)
Brief Title: Optimal Methods of Disease Progression and Survival Analysis in Children and Adults Patients With Adrenocortical Cancer (ACC)
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920095; 20-C-N095
Record Dates: First submitted 2020-04-21; First posted 2020-04-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02-10

CONDITIONS: Adrenocortical Carcinoma
Keywords: Treatment Response; Prognosis; Rare Tumor; Natural History
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Medical records of subjects enrolled on various ACC studies conducted by CCR

SUMMARY:
Background:

Adrenocortical carcinoma (ACC) is a rare cancer. It has a poor prognosis. Some people live with ACC for years; others live for just months. The average survival from the time of diagnosis is 14.5 months. Researchers do not know if local directed treatments may work better than systemic ones. They want to learn more about ACC by looking at data from previous studies.

Objective:

To characterize the overall prognosis and treatment responses in people with ACC with various systemic therapies and correlate them with age, sex, race, and disease burden.

Eligibility:

People with ACC enrolled on any of the following studies: 92-C-0268, 93-C-0200, 00-C-0044, 01-C-0129, 04-C-0011, 09-C-0242, 08-C-0176, 10-C-0203, 13-C-0114, and 14-C-0029

Design:

Study researchers will review participants medical records. They will collect the following data:

Medical record numbers

Demographics (such as age, sex, and race)

Treatments (such as surgeries, radiology procedures, and systemic treatments)

Time of disease progression between treatments and genetic/molecular data (if available)

Time of diagnosis/time of death.

All data will be kept in secure network drives or sites.

Participants who opted out of future use of data on their prior studies will be not be included in this study.

DETAILED DESCRIPTION:
Adrenocortical carcinoma (ACC) is a rare tumor with an incidence of 1.5 to 2 per million people per year. It has a very poor prognosis with an overall 5-year mortality rate of 75 - 90% and an average survival from the time of diagnosis of 14.5 months.

The natural history of ACC can vary greatly ranging from an aggressive course with patient survival measured in months to a more indolent course with patients living with the disease for years. The basis for these differing clinical presentations is not known. Therefore, accurate survival predictions in ACC are difficult and tumor classification methods with better clinical prognostic value are needed to help rationally guide the clinical management of patients with ACC. Over the last 20+ years in the CCR we have seen patients with ACC in different stages of their disease receiving various types of therapies from local directed therapies to systemic therapies, however, we have been unable to determine if local therapies may improve survival compared to the approved systemic therapies.

In this study, we plan to characterize the overall prognosis and treatment responses among patients with ACC with various systemic therapies and correlate with age, sex, race and disease burden. Identifiers will be recorded in order to correlate outcomes with therapy.

The study will involve review of patient records and will not use specimens or participant contact. The participants whose records will be reviewed in this protocol were enrolled various ACC studies conducted by CCR. The Principal Investigators of each protocol have been contacted and have given permission to conduct this study and have verified that none of the original protocols or informed consent documents precludes such a review of clinical data. Participants who did not consent to future research will be excluded.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients enrolled on any of the studies listed below:

  * 92-C-0268, 93-C-0200, 00-C-0044, 01-C-0129, 04-C-001, 09-C-0242, 08-C-0176, 10-C-0203, 13-C-0114, 14-C-0029

EXCLUSION CRITERIA:

-Patients who opted out of future use of data on their prior studies will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
response to treatment | ongoing
  prognosis and treatment responses among patients with ACC correlated with age, sex, race and disease burden

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States